CLINICAL TRIAL: NCT02258490
Title: Expanded Use of G-CSF Mobilized Donor CD34+ Selected Cells for Allogeneic Transplantation to Recipients With Limited Donor Engraftment
Brief Title: Expanded Use of G-CSF Mobilized Donor CD34+ Selected Cells for Allogeneic Transplantation
Status: No longer available | Type: Expanded Access
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Edmund Waller, Principal Investigator, Emory University
Other Study IDs: IRB00051037; EPIC-HPC001 (Other: Winship Cancer Institute)
Record Dates: First submitted 2014-09-16; First posted 2014-10-07 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Chronic Myeloid Leukemia; Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: chronic myeloid leukemia; myelodysplastic syndrome; acute myeloid leukemia; CD34+ cell mobilization therapy; graft versus host disease; allogeneic hematopoietic stem cell; G-CSF
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Graft vs Host Disease | interventions — Transplantation

INTERVENTIONS:
Biological: G-CSF mobilized CD34+ selected cells for transplantation — After screening and enrollment, donor will receive mobilization therapy with G-CSF (10 ug/Kg S/C daily x5-6 days) using standard National Marrow Donor Program guidelines. CD34+ cell selection will be performed according to procedures given in CliniMACS Operating Manual and institutional Standard Operating Procedures. If storage after CD34+ selection is necessary, product will be kept in a monitored refrigerator. During storage, leukocyte concentration should not exceed 2 x 108 cells/ml using platelet poor plasma to adjust cell concentration. If donor's plasma is not available, CliniMACS buffer will be used. Cell processing will be performed by personnel trained by Miltenyi on CliniMACS system prior to initiation of clinical product selection. After tests are performed and product passes release criteria, patient will receive final product. No conditioning regimen will be administered prior to cell infusion.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HSCT) is an established form of treatment for hematological abnormalities. Poor graft function, occurs when there poor donor engraftment. A second infusion of unselected donor hematopoietic stem cells (HSC) can result in improvement, but can potentially increase the incidence of graft versus host disease. Cluster of differentiation 34+ (CD34+) selected stem cells depleted of T-cells is an attractive alternative for treatment of poor graft function as it may be associated with less Graft versus Host Disease (GVHD) and enhanced count recovery. The investigators are using the Miltenyi CliniMACS device and CD34 cell selection reagents for the preparation of allogeneic hematopoietic progenitor cell (HPC) transplants for patients who have had prior stem cell transplants and require a stem cell "boost" from the original donor.

DETAILED DESCRIPTION:
This is a single-arm, open label, single institution, compassionate study which will enroll patients who are marginally engrafted and transfusion and/or growth factors dependent after allogeneic hematopoietic stem cell transplant (HSCT) regardless of the underlying disease for which the transplant was performed. Study subjects will receive a "booster" infusion of CD34+ cell selected and T-cell depleted G-CSF mobilized apheresis product from the original stem cell donor in order to improve engraftment. The "booster" infusion will be administered without prior conditioning.

ELIGIBILITY:
Donor Inclusion Criteria:

* Donors must be eligible and approved for a hematopoietic stem cell graft according to institutional criteria (related donor) or NMDP criteria (volunteer unrelated donor)
* Donors must be ≥ 17 years old and ≤ 75 years old
* Donors must be agreeable to receive G-CSF for CD34 cell mobilization and undergo apheresis for the second donation of peripheral blood mononuclear cells (PBMC)
* Donor must have adequate peripheral venous catheter access for apheresis or must agree to placement of a central catheter
* The following laboratory tests/evaluations will be performed for all donors registered in the study. Additional evaluations/studies may also be performed by the site as dictated by the donor's clinical situation or standard practice for monitoring normal donors

  * History and physical examination
  * Automated complete blood count (WBC, red blood cells [RBC], hematocrit, hemoglobin) with differential and platelet counts
  * Serum chemistries panel including electrolytes, glucose, blood urea nitrogen (BUN), alanine aminotransferase (ALT), creatinine, bilirubin, alkaline phosphatase, lactate dehydrogenase (LDH) and albumin. Electrolytes to include sodium, potassium, chloride, carbon dioxide, calcium and magnesium.
  * Infections disease titers by FDA licensed tests for:

    * Cytomegalovirus (CMV) antibody
    * Hepatitis panel (Hepatitis B including HBsAg, HBcAb [immunoglobulin M {IgM} and immunoglobulin G {IgG}]; hepatitis C antibody)
    * HIV 1+2 antibodies
    * Hepatitis C virus (HCV) antibodies
    * Human T-lymphotropic virus (HTLV) I/II antibodies
    * Rapid plasmin reagin (RPR)
    * HIV-1 nucleic acid amplification test (NAT)
    * HCV NAT
    * West Nile virus (WNV)
    * These tests will be obtained, and reported to Emory, within 30 days prior to collection of the CD34+ cell product.

Recipient Inclusion Criteria:

* Only patients who are experiencing life-threatening hematological insufficiency, following an allogeneic hematopoietic stem cell transplant will be enrolled into this study
* Patient must be age > 17
* Must have ≥ 90% donor cells in the unfractionated peripheral blood based on either XY fluorescence in situ hybridization (FISH) or standard short tandem repeats (STR)
* More than 60 days post allogeneic stem cell transplantation and no reversible etiology found after an allogeneic stem cell transplantation
* Must meet one of the following criteria:

  * Platelets < 20,000/μl, absolute neutrophil count (ANC) < 500/μl or
  * Transfusion dependent for at least one cell line and/or
  * On growth factor support (G-CSF) without adequate response for 30 days
* The original HSCT donor must be available, willing, and medically able to undergo G-CSF mobilization and the apheresis procedures
* Patients must have non-immune mediated graft dysfunction

Ages: 17 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Waller, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Background] Davies SM, Weisdorf DJ, Haake RJ, Kersey JH, McGlave PB, Ramsay NK, Blazar BR. Second infusion of bone marrow for treatment of graft failure after allogeneic bone marrow transplantation. Bone Marrow Transplant. 1994 Jul;14(1):73-7. PMID 7951123
- [Background] Elmaagacli AH, Peceny R, Steckel N, Trenschel R, Ottinger H, Grosse-Wilde H, Schaefer UW, Beelen DW. Outcome of transplantation of highly purified peripheral blood CD34+ cells with T-cell add-back compared with unmanipulated bone marrow or peripheral blood stem cells from HLA-identical sibling donors in patients with first chronic phase chronic myeloid leukemia. Blood. 2003 Jan 15;101(2):446-53. doi: 10.1182/blood-2002-05-1615. Epub 2002 Sep 12. PMID 12393406
- [Background] Lang P, Handgretinger R, Niethammer D, Schlegel PG, Schumm M, Greil J, Bader P, Engel C, Scheel-Walter H, Eyrich M, Klingebiel T. Transplantation of highly purified CD34+ progenitor cells from unrelated donors in pediatric leukemia. Blood. 2003 Feb 15;101(4):1630-6. doi: 10.1182/blood-2002-04-1203. Epub 2002 Oct 10. PMID 12393439
- [Background] Urbano-Ispizua A, Brunet S, Solano C, Moraleda JM, Rovira M, Zuazu J, de La Rubia J, Bargay J, Caballero D, Diez-Martin JL, Ojeda E, Perez de Oteiza JP, Ferra C, Espigado I, Alegre A, de La Serna J, Torres P, Riu C, Odriozola J, Rozman C, Sierra J, Garcia-Conde J, Montserrat E; Spanish Group of Allo-PBT. Allogeneic transplantation of CD34+-selected cells from peripheral blood in patients with myeloid malignancies in early phase: a case control comparison with unmodified peripheral blood transplantation. Bone Marrow Transplant. 2001 Aug;28(4):349-54. doi: 10.1038/sj.bmt.1703154. PMID 11571506
- [Background] Larocca A, Piaggio G, Podesta M, Pitto A, Bruno B, Di Grazia C, Gualandi F, Occhini D, Raiola AM, Dominietto A, Bregante S, Lamparelli T, Tedone E, Oneto R, Frassoni F, Van Lint MT, Pogliani E, Bacigalupo A. Boost of CD34+-selected peripheral blood cells without further conditioning in patients with poor graft function following allogeneic stem cell transplantation. Haematologica. 2006 Jul;91(7):935-40. PMID 16818281
- [Background] Tabilio A, Falzetti F, Zei T, De Ioanni M, Bonifacio E, Battelli F, Iacucci Ostini R, Ballanti S, Cimminiello M, Capponi M, Silvani C, Minelli O, Fettucciari K, Marconi P, Rosati E, Santucci A, Di Ianni M, Aversa F, Martelli MF. Graft engineering for allogeneic haploidentical stem cell transplantation. Blood Cells Mol Dis. 2004 Nov-Dec;33(3):274-80. doi: 10.1016/j.bcmd.2004.08.016. PMID 15528144
- [Background] Markiewicz M, Holowiecki J, Wojnar J, Krawczyk-Kulis M, Jagoda K, Giebel S, Kruzel T. Allogeneic transplantation of selected peripheral CD34+ cells with controlled CD3+ cells add-back in high-risk patients. Transplant Proc. 2004 Dec;36(10):3194-9. doi: 10.1016/j.transproceed.2004.09.052. PMID 15686727
- [Background] Oyekunle A, Koehl U, Schieder H, Ayuk F, Renges H, Fehse N, Zabelina T, Fehse B, Klingebiel T, Sputtek A, Zander A, Kroger N. CD34(+)-selected stem cell boost for delayed or insufficient engraftment after allogeneic stem cell transplantation. Cytotherapy. 2006;8(4):375-80. doi: 10.1080/14653240600735784. PMID 16923613
- [Background] Ringhoffer M, Wiesneth M, Harsdorf S, Schlenk RF, Schmitt A, Reinhardt PP, Moessner M, Grimminger W, Mertens T, Reske SN, Dohner H, Bunjes D. CD34 cell selection of peripheral blood progenitor cells using the CliniMACS device for allogeneic transplantation: clinical results in 102 patients. Br J Haematol. 2004 Aug;126(4):527-35. doi: 10.1111/j.1365-2141.2004.05062.x. PMID 15287946
- [Background] Kao GS, Kim HT, Daley H, Ritz J, Burger SR, Kelley L, Vierra-Green C, Flesch S, Spellman S, Miller J, Confer D. Validation of short-term handling and storage conditions for marrow and peripheral blood stem cell products. Transfusion. 2011 Jan;51(1):137-47. doi: 10.1111/j.1537-2995.2010.02758.x. PMID 20609197
- [Background] Antonenas V, Garvin F, Webb M, Sartor M, Bradstock KF, Gottlieb D. Fresh PBSC harvests, but not BM, show temperature-related loss of CD34 viability during storage and transport. Cytotherapy. 2006;8(2):158-65. doi: 10.1080/14653240600620994. PMID 16698689